CLINICAL TRIAL: NCT01666665
Title: Mechanisms of Improved Wound Healing and Protein Synthesis of Insulin and Metformin
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: At the request of the study site, this study has been closed and access to study-related data is unavailable. We are unable to submit the results-data.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 12-142
Record Dates: First submitted 2012-08-06; First posted 2012-08-16 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2018-08

CONDITIONS: Insulin Resistance; Hypermetabolism; Hyperglycemia
Keywords: Burn
MeSH Terms: conditions — Insulin Resistance; Hyperglycemia; Burns | interventions — Metformin; Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformin (Active Comparator): Metformin up to 1000mg/m2 body surface area by mouth of feeding tube up to 3 times each day for 12 months
  Interventions: Drug: Metformin
- Sugar pill (Placebo Comparator): sugar pill up to 3 times per day for 12 months
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Metformin — Metformin up to 1000mg/m2 body surface area by mouth of feeding tube up to 3 times each day for 12 months
  Other Names: glucophage
  Arms: metformin
Drug: Sugar pill — Sugar pill up to 3 times per day for 12 months
  Other Names: placebo
  Arms: Sugar pill

SUMMARY:
Massive pediatric burns are associated with a persistent and sustained hypermetabolic response characterized by elevated levels of circulating catecholamine's, cortisol, and glucagon's, which can cause extreme muscle wasting, immunodeficiency, and delay in wound healing. Insulin and metformin have demonstrated anabolic activity with minimal associated side effects. However, it is unknown whether the beneficial effects arise from tight euglycemic control or direct effect of insulin action. We hypothesize that during acute hospitalization, administration of metformin at a dose titrated to maintain blood glucose between 80-180 mg/dl will accelerate wound healing and recovery in children with severe thermal injury and will have beneficial long-term effects on muscle strength, immune function, and wound healing.

DETAILED DESCRIPTION:
Metformin treated patients will be compared to control patients. Both groups will receive insulin therapy for blood glucose >180mg/dl. Insulin will be titrated according to hospital sliding scale.

The use of insulin or metformin will benefit burned children by improving muscle protein build-up, speeding wound healing and reversing growth arrest, improving the immune response, and positively affecting long-term rehabilitation.

The results of this study may initiate a change in standard of care as it is found that simply the reduction of blood glucose by metformin, improves patient outcomes as metformin can be administered without the added complication of hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 10-19
* Primary diagnosis of ≥ 20 Total Burn Surface Area Burn (TBSAB )

Exclusion Criteria:

* Decision not to treat due to burn injury severity
* Known history of AIDS, ARC, HIV
* Pregnancy
* Previous diagnosis (pre -burn) of renal failure, liver disease or hepatic dysfunction- Serum Creatinine >1.5mg/dL for males and >1.4mg/dL for females, after fluid resuscitation (Clinical definition of kidney damage)
* Pre-existing type 1 diabetes mellitus
* Pre Existing type 2 diabetes mellitus and receiving treatment
* Allergies to Metformin
* Acute or chronic acidosis (lactic or any other metabolic type) and renal failure

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | Measure changes between admission and 2 years post burn
  As measured by OGTT

SECONDARY OUTCOMES:
Protein synthesis | Measure changes between admission and 1 years post burn
  As measured by stable isotope infusion study
Morbidity | Measure changes between admission and 2 years post burn
  As measured by Organ Failure assessments

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — University of Texas
Locations (1):
- Shriners Hospitals for Children, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No